CLINICAL TRIAL: NCT07223853
Title: Intelligent Clinical Decision Support for Preoperative Blood Management: A Cluster-Randomized Clinical Trial
Brief Title: AI-driven Clinical Decision Support for Perioperative Blood Orders
Acronym: SPATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sunny Lou, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 202506199; K23HL166880 (NIH)
Record Dates: First submitted 2025-10-28; First posted 2025-11-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Surgery
Keywords: artificial intelligence; clinical decision support; machine learning; surgery; perioperative blood management; anesthesia; pretransfusion testing

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care for determining presurgical blood orders, including use of the institutional Maximum Surgical Blood Ordering Schedule (MSBOS)
  Interventions: Other: Usual care
- S-PATH (Experimental): Access to the S-PATH clinical decision support system
  Interventions: Other: S-PATH clinical decision support system

INTERVENTIONS:
Other: S-PATH clinical decision support system — Access to the S-PATH electronic health record (EHR)-integrated clinical decision support system
  Arms: S-PATH
Other: Usual care — Including use of the conventional Maximum Surgical Blood Ordering Schedule (MSBOS)
  Arms: Usual care

SUMMARY:
20 million patients have surgery in the United States every year, with approximately 1 million of those patients requiring life-saving blood transfusion. Presurgical preparation for transfusion is important to allow for safe and timely transfusion during surgery; however, excessive preparation is unfortunately common, costly, and contributes to blood waste. This study aims to evaluate an intelligent clinical decision support system that helps clinicians prepare blood for patients who are likely to need it, while avoiding excessive preparation for patients who don't, potentially improving patient safety while reducing blood waste and healthcare costs.

ELIGIBILITY:
Clinician Level Exclusion Criteria:

* Clinician (resident physician or advanced practice provider) who works at a preoperative assessment clinic

Clinician Level Exclusion Criteria:

* None

Patient Inclusion Criteria:

* Scheduled for surgery in one of the main operating room areas (non-remote) at Barnes Jewish Hospital
* Evaluated in-person at one of the preoperative assessment clinics affiliated with BJC Healthcare
* Have a valid S-PATH model prediction prior to their preoperative assessment clinic visit

Patient Exclusion Criteria:

* Pregnant
* Presence or history of red cell alloantibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with a type and screen order placed during the preoperative clinic assessment visit | Decision made during the preoperative assessment clinic visit
  This is a binary outcome at the patient / surgical case level, which will be aggregated across all patients in the study to produce an overall frequency. Placement of a type and screen order during the preoperative clinic assessment visit will be evaluated at the patient / surgical case level. This includes orders placed and collected during the preoperative clinic assessment visit, as well as orders signed during the preoperative clinic assessment visit or subsequent follow up care and held to be drawn on the day of surgery.

SECONDARY OUTCOMES:
Frequency of a valid type and screen order at the start of surgery | Start of surgery (1 hour after Anesthesia Start)
  This is a binary outcome at the patient / surgical case level, which will be aggregated across all patients in the study to produce an overall frequency. Valid type and screen order at the start of surgery (defined as resulted prior to 1h after anesthesia start). The 1 hour buffer is used to account for orders that were drawn prior to surgery but may not have resulted by the time the patient enters the operating room. This will include orders placed by the clinicians working in preoperative assessment clinic and any orders that may be placed by the day of surgery anesthesia or surgical teams. This will not include type and screen orders that have expired by the start of surgery. This is a secondary efficacy outcome that reflects type and screen ordering decisions by all members of the patient's care team.
Frequency of red cell transfusion during surgery | During surgery
  This is a binary outcome at the patient / surgical case level, which will be aggregated across all patients in the study to produce an overall frequency. Administration of allogeneic packed red blood cells during surgery will be retrieved from the electronic health record. Documentation of transfusion is mandatory and the electronic health record scan is used to confirm the correct patient. This is a secondary efficacy outcome, as lack of a type and screen may prevent discretionary intraoperative transfusion.
Frequency of emergency release blood use during surgery | During surgery
  This is a binary outcome at the patient / surgical case level, which will be aggregated across all patients in the study to produce an overall frequency. Administration of emergency release allogeneic packed red blood cells will be retrieved from the electronic health record. These are either documented as volumes under the MTP tab or individually scanned as uncrossmatched red cells. This is the primary safety outcome of the study as emergency release blood may be administered if red cell transfusion is urgently indicated but a type and screen is not available. The frequency of this outcome will be reported overall across both groups, and stratified by whether the patient had an active type and screen at the start of surgery.
Frequency of red cell transfusion during surgery without an active type and screen at the start of surgery | During surgery
  This is a binary outcome at the patient / surgical case level, which will be aggregated across all patients in the study to produce an overall frequency. This is the secondary safety outcome intended to capture false negative results, i.e., patients who required transfusion during surgery but did not have a preoperative type and screen. This outcome will be collected electronically from the EHR and will capture patients for whom the type and screen was resulted after the start of surgery (i.e., after 1h after anesthesia start), suggesting it was collected after the patient entered the operating room
Frequency of transfusion reaction | From time of surgery to hospital discharge or 30 days after surgery
  This is a binary outcome at the patient / surgical case level, which will be aggregated across all patients in the study to produce an overall frequency. Transfusion reactions are reported by clinical teams to the blood bank, and the transfusion medicine service investigates and classifies each transfusion reaction. These investigation reports will be transmitted to the study team for adverse event reporting and outcome collection. This is also a secondary safety outcome for the study. Transfusion reactions will be reported stratified by category, as hemolytic transfusion reactions are the most relevant to the trial.

OTHER OUTCOMES:
Viewing S-PATH predictions (Implementation outcome) | Through study completion, an average of 1 year
  Clinician-level measure of the frequency of viewing S-PATH predictions, retrieved from EHR audit log data
Acceptance of S-PATH recommendation (Implementation outcome) | Through study completion, an average of 1 year
  Clinician-level measure of the frequency of the clinician's blood order during the preoperative clinic visit (1' outcome) matching S-PATH's recommendation
Cost assessment | Through study completion, an average of 1 year
  Estimate of the cost savings associated with S-PATH use

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University / Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
For each clinician, the final dataset will include self-reported demographic information, exit interview transcripts, and behavioral and implementation outcomes relating to usage of the proposed clinical decision support (CDS) intervention.
  For each patient, the final dataset will include clinical and safety outcomes for the study.
  Trial materials, including consent forms, protocols, and code book for qualitative analysis will also be shared.
  To anonymize the data, all clinicians and patients will be assigned random identifiers to replace clinician names and patient medical record numbers. No dates for surgical encounters will be retained. All other incidental identifiers (such as mentions of care team member names, encounter numbers, or hospital units) will be stripped.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available within 12 months of the grant period ending or on publication of a manuscript using the data, whichever comes first. Data will be retained in the WashU Libraries Open Scholarship Digital Research Materials Repository for at least 10 years.
Access Criteria: The proposed clinical trial will involve a near-complete sampling of clinicians who work at the host institution's preoperative assessment clinic. Even with removal of identifiers, we believe it would be difficult to protect the identities of clinician participants given the type of demographic data collected and the very restricted setting in which recruitment will occur. In addition, even if patient data is anonymized, it may be possible to reidentify the patients using metadata alone. Therefore, access controls will be required prior to sharing of the all data, including patient and clinician data. Specifically, data will be shared only under a data-sharing agreement according to institutional guidelines that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are complete.

REFERENCES:
- [Background] Yang P, Zijlstra EP, Hall BL, Gregory SH, Jackups R Jr, Li J, Abraham J, Lou SS. Challenges in reliable preoperative blood ordering: A qualitative interview study. Transfusion. 2024 Oct;64(10):1889-1898. doi: 10.1111/trf.18012. Epub 2024 Sep 16. PMID 39279676
- [Background] Lou SS, Liu H, Lu C, Wildes TS, Hall BL, Kannampallil T. Personalized Surgical Transfusion Risk Prediction Using Machine Learning to Guide Preoperative Type and Screen Orders. Anesthesiology. 2022 Jul 1;137(1):55-66. doi: 10.1097/ALN.0000000000004139. PMID 35147666
- [Background] Lou SS, Liu Y, Cohen ME, Ko CY, Hall BL, Kannampallil T. National Multi-Institutional Validation of a Surgical Transfusion Risk Prediction Model. J Am Coll Surg. 2024 Jan 1;238(1):99-105. doi: 10.1097/XCS.0000000000000874. Epub 2023 Sep 22. PMID 37737660
- [Background] Lou SS, Kumar S, Goss CW, Avidan MS, Kheterpal S, Kannampallil T; Multicenter Perioperative Outcomes Group. Multicenter Validation of a Machine Learning Model for Surgical Transfusion Risk at 45 US Hospitals. JAMA Netw Open. 2025 Jun 2;8(6):e2517760. doi: 10.1001/jamanetworkopen.2025.17760. PMID 40577014

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT07223853/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT07223853/ICF_001.pdf